CLINICAL TRIAL: NCT00900952
Title: Epidemiologic Study of Infections in Elderly Patients
Brief Title: Epidemiologic Study Evaluating Infections in Elderly Patients
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Other Study IDs: 3074X1-4489
Record Dates: First submitted 2009-05-07; First posted 2009-05-13 (Estimated); Last update posted 2009-10-09 (Estimated); Status verified 2009-10

CONDITIONS: Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Infected elderly patients
  Interventions: Other: Clinical record review

INTERVENTIONS:
Other: Clinical record review

SUMMARY:
The purpose of this observational study is to assess the prevalence and demographic and clinical characteristics of infections in elderly people admitted to Internal Medicine wards in Spain, as well as the etiology and resistance pattern for the main causal agents, and outcome.

ELIGIBILITY:
Inclusion criteria:

* Patients > 65 years of age that are hospitalized in an Internal Medicine ward and have an active infection (skin and soft tissue, intra-abdominal, or respiratory infections) from the community that needs antibiotic treatment
* Patients must have at least one sample processed for microbiological diagnosis

Exclusion criteria:

* COPD exacerbation
* Urinary tract infections
* Hospital acquired infections
* Other infections not in inclusion criteria

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Infected elderly patients treated at Internal Medicine wards in Spanish hospitals
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of each kind of infection will be measured from a descriptive point of view, using relative and absolute frequencies. | 5 months

SECONDARY OUTCOMES:
Study the etiology and resistance pattern for the main causal agents. | 5 months
Describe the demographic features, co-morbidities, concomitant treatment and outcome of patients. | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Mataró, Barcelona, Spain